CLINICAL TRIAL: NCT05197998
Title: Promoting ColorBRAVE Conversations in Families: A Public Health Strategy to Advance Racial Equity
Brief Title: Promoting ColorBRAVE Conversations in Families
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Early Termination of Grant
Sponsor: Tulane University (Other)
Collaborators: Tufts University (Other); University of Chicago (Other); University of Illinois at Chicago (Other); San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1U01OD033242-01 (NIH)
Record Dates: First submitted 2021-11-22; First posted 2022-01-20 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Child Development; Parents; Prosocial and Emotional Well-Being

STUDY DESIGN:
Intervention Model Description: Wait-list control design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ColorBRAVE (Experimental): The experimental group will be asked to download a multi-module mobile app designed to guide parents and caregivers in having conversations about race with their K-2nd grade children
  Interventions: Behavioral: ColorBRAVE
- Wait-list Control (Other): The wait-list control group will be placed on the wait-list for the first 6-weeks, the period in which the experimental group will complete the intervention program. Following the 6-week wait-list period they will receive the ColorBRAVE program.
  Interventions: Behavioral: ColorBRAVE

INTERVENTIONS:
Behavioral: ColorBRAVE — The intervention is a multi-module program delivered via a mobile app for parents of children in K-2nd grade. Each module in the program will take approximately 30 minutes to complete, with lessons facilitated through interactive storytelling, videos, and games.

SUMMARY:
The objective of this research is to evaluate a mobile app-based intervention for parents of children in K-2nd grade designed that guides them in how to have productive conversations about race with their children. This study will recruit a national sample of parents and their K-2nd grade children. The impact of the intervention is tested using a wait-list controlled trial design. Outcomes include prosocial behaviors and indicators of emotional well-being.

ELIGIBILITY:
Residence in the US; caregiver age 18 years or older and child age 5-8 years old; ability to read and understand English

Ages: 5 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Racial Socialization Frequency Scale | 0-12 months
  Parents will report the frequency with which they engage in racial socialization practices with their K-2nd grade child.
Racial Socialization Competency Scale | 0-12 months
  Parents will report the degree of comfort, skills, and stress in engaging in different processes related to racial socialization with their K-2nd grade child.
Cross-race Friendships | 0-12 months
  Parents will report the race of their K-2nd grade child's 5 closest friends - the number of cross-race friendships will consist of the number of friends that are race discordant to their child.
Colorblind Racial Attitudes (CoBRAS) Scale | 0-12 months
  Color-blind racial attitudes among parents will be assessed using the COBRAS Scale.
Child Prosocial Behavior Questionnaire (CPBQ) | 0-12 months
  Parents will report on the degree to which their K-2nd grade child engages in various prosocial behaviors, including those surrounding helping, sharing, and comforting.
Patient-Reported Outcomes Measurement Information System (PROMIS) Parent Proxy Measures | 0-12 months
  Parent reports of child socio-emotional well being (e.g., positive peer relationships, depression, anxiety).
Prosocial Children Measure | 0-12 months
  Children (ages 5-8 years old) will be introduced to a child and told scenarios in which that child must choose other children to engage in various activities with, among a group of diverse children. Children will be asked (1) whether they liked or disliked how that child chose the children to participate in the activity with and (2) if there is anything they would like to say to that child about their choice in children.
Child Bystander Response Questionnaire | 0-12 months
  Children will report the frequency with which they engage in different bystander behaviors when they see someone being treated poorly or unfairly due to their race, ethnicity, or cultural background.

CONTACTS AND LOCATIONS:
Overall Officials: David H. Chae, ScD, MA, Principal Investigator — Tulane University
Locations (1):
- Tulane University, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of key analyses, study documentation and de-identified data will be made available to the research community upon request. Data requests may be submitted to the Project Coordinator and reviewed by the study PI to determine whether there is significant scientific overlap in the research questions and analyses proposed by the outside investigator. Those who submit qualified proposals will be provided with a dataset containing only the variables requested and the associated documentation (e.g., codebooks, description of study protocols, data dictionaries) under a data sharing agreement.